CLINICAL TRIAL: NCT00740090
Title: Phase 1, Randomized, Double-Blind, Dose-Escalating Study of the Safety, Reactogenicity, and Immunogenicity of the AMA1-C1/Alhydrogel+CPG 7909 Vaccine for Plasmodium Falciparum Malaria in Children in Mali
Brief Title: Malaria Vaccine for Children in Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 999908194; 08-I-N194
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-06-09

CONDITIONS: Malaria; Malaria Infection
Keywords: Malaria; Reactogenicity, Safety, Immunogenicity; Maleria Endemic; Plasmodium Falciparum; Dose Escalating
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — ProMune

INTERVENTIONS:
Drug: AMA1-C1/Alhydrogel plus CPG 7909

SUMMARY:
This study will evaluate the safety and immune response of children to an experimental malaria vaccine called AMA1-C1/Alhydrogel® (Registered Trademark) + CPG 7909. Malaria is an infection of red blood cells caused by a parasite, Plasmodium falciparum, that is spread by certain kinds of mosquitoes. It affects at least 300 million people worldwide each year, with more than 1 million deaths, mostly among children less than 5 years of age in sub-Saharan Africa. Malaria is the leading cause of death and illness among the general population of Mali in West Africa. Increasing drug resistance to P. falciparum and widespread resistance of mosquitoes to pesticides are reducing the ability to control the disease through these strategies. AMA1 C1 is made from a synthetic protein similar to a P. falciparum protein. It is combined with Alhydrogel and CPG 7909, substances added to vaccines to make them work better.

Children between 1 and 4 years of age who live in Bancoumana, Mali, and are in general good health may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood and urine tests.

Participants are randomly assigned to receive three injections (shots) of either AMA1-C1 or a control rabies inactivated vaccine called Imovax® (Registered Trademark). The shots are given in the thigh muscle on study days 0, 56 and 180. After each shot, participants are observed in the clinic for 30 minutes. They return to the clinic for a physical examination six or seven times between each shot and then four more times over a 9-month period after the last shot. Blood samples are drawn at several of these visits to check for side effects of the vaccine and to measure the response to it. The total duration of the study is 21 months.

...

DETAILED DESCRIPTION:
Globally, the Plasmodium falciparum parasite is responsible for at least 300 million acute cases of malaria each year, with more than 1 million deaths. Approximately 90 percent of these deaths, the majority in children under 5 years of age, occur in Africa due to infection with Plasmodium falciparum. Morbidity and mortality caused by malaria also has significant direct and indirect costs on the economic development of the endemic countries. It is estimated that malaria accounts for 40 percent of public health expenditures, more than 30 percent of inpatient admissions, and approximately 50 percent of outpatient visits in some African countries. These factors, as well as growing drug resistance of the parasite, widespread resistance of mosquitoes to insecticide, and increased human travel necessitate the need for new approaches to malaria control and eradication. A vaccine that could reduce both mortality and morbidity secondary to Plasmodium falciparum infection would be a valuable resource in the fight against this disease.

Over time, people living in endemic areas develop natural immunity to Plasmodium falciparum as a result of repeated infection. Consequently, children who survive to 7 to 10 years of age rarely succumb to life-threatening disease despite frequent infection. This acquired immunity is mediated in part by blood-stage parasite-specific antibodies. Thus, parasite proteins expressed during the blood-stage have been proposed to be good candidates for inclusion in a vaccine. The purpose of a blood-stage vaccine is to elicit immune responses that either destroy the parasite in the blood stream or inhibit the parasite from infecting red blood cells, thus reducing or preventing complications of the disease.

A number of Plasmodium falciparum merozoite antigens have been identified as promising blood-stage vaccine candidates, including Apical Membrane Antigen 1 (AMA1). The precise role of AMA1 in the parasite is unknown; however, it is critical in the erythrocyte invasion process across divergent Plasmodium species and for blood-stage multiplication of the parasite. Recent analysis of the Plasmodium falciparum proteome detected expression of AMA1 in the sporozoite stage and suggests an additional role for AMA1 during the liver-stage invasion. Therefore, an immune response against AMA1 may have an effect on liver-stage parasites as well as having an impact on blood-stage parasites, thus protecting the host by multiple immune mechanisms. Human and animal anti-AMA1 antibodies inhibit merozoite invasion in vitro and correlate with protection against parasite challenge in animal models. T-cells specific for Plasmodium falciparum AMA1 have also been demonstrated in individuals living in endemic areas.

At least 68 known amino acid polymorphisms of AMA1 have been demonstrated, and animal studies have shown that the polymorphisms in AMA1 are not immunologically silent. The combination of two or more divergent AMA1 sequences within a single vaccine formulation may reduce evasion of the host immune response by some Plasmodium falciparum field isolates.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males or females aged greater than or equal to 1 to less than 4 years

Known residents of the village of Bancoumana, Mali or its surrounding area

Good general health as determined by means of the screening procedure

Available for the duration of the trial (24 months from enrollment)

Willingness to have child participate in the study as evidenced by parents/legal guardians signing or fingerprinting the informed consent document

EXCLUSION CRITERIA:

Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, chronic infectious or renal disease by history, physical examination, and/or laboratory studies including urinalysis.

Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer or the parent/legal guardian to understand and cooperate with the study protocol.

Pre-existing known autoimmune diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, or autoimmune thrombocytopenia.

Laboratory evidence of possible autoimmune disease determined by anti-dsDNA titer that equals or exceeds 25 IU.

Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than the upper limit of normal of the testing laboratory).

Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory, or more than trace protein or blood on urine dipstick testing confirmed by repeat testing).

Laboratory evidence of hematologic disease (absolute leukocyte count less than 3000/mm(3) or greater than 14,500/mm(3), absolute lymphocyte count less than 1000/mm(3), platelet count less than 120,000/mm(3), or hemoglobin less than 8.5 g/dL).

Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Participation in another investigational vaccine or drug trial within 30 days of starting this study, or while this study is ongoing.

History of a severe allergic reaction or anaphylaxis.

History of allergy to nickel.

Severe asthma. This will be defined as:

Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or parenteral corticosteroids.

Clinically significant reactive airway disease that does not respond to bronchodilators.

Positive screening test for anti-Hepatitis C virus (anti-HCV).

Positive screening test for Hepatitis B surface antigen (HBsAg).

Known immunodeficiency syndrome.

Use of systemic corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study.

History of a surgical splenectomy.

Receipt of blood products within the past 6 months.

Previous receipt of an investigational malaria vaccine or of rabies vaccine.

History of use of chloroquine or related compounds (amodiaquine or primaquine) within 8 weeks of study entry. Chloroquine and related compounds have the potential to interfere with CPG-induced activation of B cells and plasma dendritic cells.

Previous administration of Verorab Trademark vaccine.

Known thrombocytopenia or bleeding disorders.

Known allergy to neomycin (a component of Verorab Trademark).

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200
Dates: Start 2008-08-11; Primary Completion 2009-06-09 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of systemic and local adverse events.

SECONDARY OUTCOMES:
Antibody response determined by ELISA, to the AMA1-FVO and AMA1-3D7 proteins at selected time points. Inhibition of P. falciparum FVO and 3D7 parasite growth in vitro determined at selected time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Sachs J, Malaney P. The economic and social burden of malaria. Nature. 2002 Feb 7;415(6872):680-5. doi: 10.1038/415680a. PMID 11832956
- [Background] Richie TL, Saul A. Progress and challenges for malaria vaccines. Nature. 2002 Feb 7;415(6872):694-701. doi: 10.1038/415694a. PMID 11832958
- [Background] Triglia T, Healer J, Caruana SR, Hodder AN, Anders RF, Crabb BS, Cowman AF. Apical membrane antigen 1 plays a central role in erythrocyte invasion by Plasmodium species. Mol Microbiol. 2000 Nov;38(4):706-18. doi: 10.1046/j.1365-2958.2000.02175.x. PMID 11115107